CLINICAL TRIAL: NCT02986568
Title: Cohort Study for Comparing the Efficacy Between the Standard Treatment and Fusion Ontogenetic Surgery for Gynecologic Cancers (FUSION Trial IV)
Brief Title: Efficacy of the Standard Treatment and Fusion Ontogenetic Surgery for Gynecologic Cancers
Acronym: FUSIONIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee Seung Kim, Associate Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-1616
Record Dates: First submitted 2016-10-16; First posted 2016-12-08 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Cervical Cancer; Uterine Cancer
Keywords: Ontogenetic surgery; TMMR; PMMR; LEER
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cervical cancer (Experimental): * Primary cervical cancer patients, FIGO stage IB1-IIB
  * Refractory cervical cancer patients who do not respond to concurrent chemoradiotherapy or radiotherapy
  * Recurrent cervical cancer after concurrent chemoradiotherapy or radiotherapy
  Interventions: Procedure: Cervical cancer
- Uterine cancer (Experimental): * Primary uterine cancer patients, FIGO stage IA, grade3, IB-IVA
  * Refractory uterine cancer who does not respond to concurrent chemoradiotherapy or radiotherapy
  * Recurrent uterine cancer after concurrent chemoradiotherapy or radiotherapy
  Interventions: Procedure: Uterine cancer
- Cervical cancer, pelvic sidewall invasion (Experimental): Cervical cancer patients showing pelvic sidewall invasion
  * Primary cervical cancer
  * Refractory cervical cancer patients who do not respond to concurrent chemoradiotherapy or radiotherapy
  * Recurrent cervical cancer after concurrent chemoradiotherapy or radiotherapy
  Interventions: Procedure: Cervical cancer, pelvic sidewall invasion
- Non-cervical cancer, pelvic sidewall invasion (Experimental): * Gynecologic cancer patients other than cerivcal cancer, showing pelvic sidewall invasion with or without distant metastasis
  * Patients showing uncontrolled pelvic pain due to the tumor invasion
  Interventions: Procedure: Non-cervical cancer, pelvic sidewall invasion

INTERVENTIONS:
Procedure: Cervical cancer — If tumor sized ≥ 5cm, undergo neoadjuvant chemotherapy with Cisplatin before surgery. (40mg/m2 on day 1 of each 7 day cycle for 5 cycles), then perform Fusion TMMR after neoadjuvant chemotherapy with cisplatin as above.
  If tumor size < 5cm, perform Fusion Total mesometrial resection (TMMR)
  After surgery, if resection margin, more than two pelvic lymph node or more than one para-aortic lymph node is positive in pathologic report, undergo adjuvant chemotherapy.
  If not, no adjuvant therapy.
  Arms: Cervical cancer
Procedure: Uterine cancer — Perform Fusion Peritoneal mesometrial resection (PMMR).
  After surgery, if resection margin, more than two pelvic lymph node or more than one para-aortic lymph node is positive in pathologic report, undergo adjuvant chemotherapy.
  If not, no adjuvant therapy.
  Arms: Uterine cancer
Procedure: Cervical cancer, pelvic sidewall invasion — Perform Fusion Laterally extended endopelvic resection (LEER).
  After surgery, if resection margin, more than two pelvic lymph node or more than one para-aortic lymph node is positive in pathologic report, undergo adjuvant chemotherapy. Patients with primary disease will be treated with adjvuant chemotherapy. In case of recurrent disease, bevacizumab, paclitaxel, and cisplaitn will be administered regardless of the pathologic report (bevacizumab 15mg/kg on day 1, paclitaxel 135mg/m2 on day 1, and cisplatin 50mg/m2 on day 2, of each 21 day cycle).
  If not, no adjuvant therapy.
  Arms: Cervical cancer, pelvic sidewall invasion
Procedure: Non-cervical cancer, pelvic sidewall invasion — Perform Fusion Laterally extended endopelvic resection (LEER).
  After surgery, appropriate adjuvant chemotherapy will be administered depending on the tumor type.
  Arms: Non-cervical cancer, pelvic sidewall invasion

SUMMARY:
The purpose of this study is to compare standard treatment and fusion ontogenetic surgery (total mesometrial resection, laterally extended endopelvic resection, peritoneal mesometrial resection) for gynecologic cancer in order to evaluate treatment response, adverse effect and survival.

DETAILED DESCRIPTION:
Fujii method and ontogenetic surgery are the surgical method of radical hysterectomy that can preserve pelvic organ function as much as possible.

Fujii method has advantage of preserving pelvic autonomic nerve with radical resection of tissue under parametrium. And ontogenetic surgery has advantage of reducing need of radiation therapy by radical resection of tissue above parametrium.

This study is prospective study for fusion ontogenetic surgery that has the advantage of both Fujji method and ontogenetic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female, Age ≥ 20 years
* Patients with primary, recurrent, or refractory cervical cancer (FIGO stage IB1-IVA), primary, recurrent, or refractory uterine cancer (FIGO stage IA, grade 3, IB-IVA), or gynecologic cancer patients showing pelvic sidewall recurrence.
* ECOG performance status 0 or 1
* Extensive surgery might be expected to cure the disease, or expected to relieve severe pelvic pain.
* Patients who signed an approved informed consent
* Patients who do not have a treatment option other than surgery.

Exclusion Criteria:

* Female, Age < 20 years
* ECOG performance status ≥2
* Bilateral pelvic sidewall invasion
* Patients who had undergone radical hysterectomy, trachelectomy, or hysterectomy in case of the primary disease.
* Patients who refused to sign an informed consent

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2016-05-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From date of treatment start until the date of first documented progression or date of death (by any cause, in the absence of disease progression) whichever came first, assessed up to 60 months
  The time interval from treatment start date to disease recurrence or progression date
Overall survival | From the date of treatment start until death due to any cause, assessed up to 60 months
  the time interval from treatment start date to death or end of study date
Treatment-free interval | From date of treatment end until the date of first documented progression or date of death (by any cause, in the absence of disease progression) whichever came first, assessed up to 60 months
  The time interval from treatment end date to disease recurrence or progression date
Treatment-related survival | the time interval from treatment start date to death or end of study date assessed up to 60 months
  the time interval from treatment start date to death or end of study date (recurrent or refractory disease)

SECONDARY OUTCOMES:
Tumor response | 3 weeks after completion of ontogenetic surgery up to 6 weeks
  Tumor response after surgery, and the evaluation is based on revised RECIST version 1.1
Postoperative complications 1 | after the ontogenetic surgery, up to 30 days
  Incidence of early complications, and severity of complications based on Memorial Sloan Kettering Cancer Center Surgical Secondary Events Grading System
Postoperative complications 2 | 31 days after the ontogenetic surgery through study completion, an average of 1 year
  Incidence of late complications, and severity of complications based on Memorial Sloan Kettering Cancer Center Surgical Secondary Events Grading System
Neurologic disturbance of low extremity | after the ontogenetic surgery, up to 30 days
  Incidence of motor and sensory disturbances of low extremities, and the grading is based on Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Pain evaluation | 1 day before the ontogenetic surgery, and at the time of discharge after postoperative management of the ontogenetic surgery assessed up to 60 months
  Pelvic pain evaluated by numeric rating scale and morphine milligram equivalents (MME)
Time to normal bladder function | The time from the ontogentic surgery to the time of confirmation or normal bladder function, assessed up to 60 months
  In case of bladder preservation, normal bladder function is evaluated by residual urine check after time voiding, and the volume of residual urine is less than 100cc.
  The time from the ontogentic surgery to the time of confirmation or normal bladder function.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Seung Kim, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piver MS, Rutledge F, Smith JP. Five classes of extended hysterectomy for women with cervical cancer. Obstet Gynecol. 1974 Aug;44(2):265-72. No abstract available. PMID 4417035
- [Background] Querleu D, Morrow CP. Classification of radical hysterectomy. Lancet Oncol. 2008 Mar;9(3):297-303. doi: 10.1016/S1470-2045(08)70074-3. PMID 18308255
- [Background] Koh WJ, Greer BE, Abu-Rustum NR, Apte SM, Campos SM, Cho KR, Chu C, Cohn D, Crispens MA, Dorigo O, Eifel PJ, Fisher CM, Frederick P, Gaffney DK, Han E, Huh WK, Lurain JR 3rd, Mutch D, Fader AN, Remmenga SW, Reynolds RK, Teng N, Tillmanns T, Valea FA, Yashar CM, McMillian NR, Scavone JL. Cervical Cancer, Version 2.2015. J Natl Compr Canc Netw. 2015 Apr;13(4):395-404; quiz 404. doi: 10.6004/jnccn.2015.0055. PMID 25870376
- [Background] Koh WJ, Greer BE, Abu-Rustum NR, Apte SM, Campos SM, Chan J, Cho KR, Cohn D, Crispens MA, Dupont N, Eifel PJ, Fader AN, Fisher CM, Gaffney DK, George S, Han E, Huh WK, Lurain JR 3rd, Martin L, Mutch D, Remmenga SW, Reynolds RK, Small W Jr, Teng N, Tillmanns T, Valea FA, McMillian N, Hughes M. Uterine neoplasms, version 1.2014. J Natl Compr Canc Netw. 2014 Feb;12(2):248-80. doi: 10.6004/jnccn.2014.0025. PMID 24586086
- [Background] Fujii S. Anatomic identification of nerve-sparing radical hysterectomy: a step-by-step procedure. Gynecol Oncol. 2008 Nov;111(2 Suppl):S33-41. doi: 10.1016/j.ygyno.2008.07.026. Epub 2008 Aug 27. PMID 18752840
- [Background] Kim HS, Kim TH, Suh DH, Kim SY, Kim MA, Jeong CW, Hong KS, Song YS. Success Factors of Laparoscopic Nerve-sparing Radical Hysterectomy for Preserving Bladder Function in Patients with Cervical Cancer: A Protocol-Based Prospective Cohort Study. Ann Surg Oncol. 2015;22(6):1987-95. doi: 10.1245/s10434-014-4197-1. Epub 2014 Dec 3. PMID 25465377
- [Background] Kim HS, Kim K, Ryoo SB, Seo JH, Kim SY, Park JW, Kim MA, Hong KS, Jeong CW, Song YS; FUSION Study Group. Conventional versus nerve-sparing radical surgery for cervical cancer: a meta-analysis. J Gynecol Oncol. 2015 Apr;26(2):100-10. doi: 10.3802/jgo.2015.26.2.100. PMID 25872891
- [Background] Hockel M, Horn LC, Fritsch H. Association between the mesenchymal compartment of uterovaginal organogenesis and local tumour spread in stage IB-IIB cervical carcinoma: a prospective study. Lancet Oncol. 2005 Oct;6(10):751-6. doi: 10.1016/S1470-2045(05)70324-7. Epub 2005 Sep 8. PMID 16198980
- [Background] Hockel M. Laterally extended endopelvic resection. Novel surgical treatment of locally recurrent cervical carcinoma involving the pelvic side wall. Gynecol Oncol. 2003 Nov;91(2):369-77. doi: 10.1016/s0090-8258(03)00502-x. PMID 14599868
- [Background] Hockel M, Horn LC, Einenkel J. (Laterally) extended endopelvic resection: surgical treatment of locally advanced and recurrent cancer of the uterine cervix and vagina based on ontogenetic anatomy. Gynecol Oncol. 2012 Nov;127(2):297-302. doi: 10.1016/j.ygyno.2012.07.120. Epub 2012 Aug 1. PMID 22864112
- [Background] Hockel M, Horn LC, Manthey N, Braumann UD, Wolf U, Teichmann G, Frauenschlager K, Dornhofer N, Einenkel J. Resection of the embryologically defined uterovaginal (Mullerian) compartment and pelvic control in patients with cervical cancer: a prospective analysis. Lancet Oncol. 2009 Jul;10(7):683-92. doi: 10.1016/S1470-2045(09)70100-7. Epub 2009 May 29. PMID 19482513
- [Background] Hockel M, Hentschel B, Horn LC. Association between developmental steps in the organogenesis of the uterine cervix and locoregional progression of cervical cancer: a prospective clinicopathological analysis. Lancet Oncol. 2014 Apr;15(4):445-56. doi: 10.1016/S1470-2045(14)70060-9. Epub 2014 Mar 19. PMID 24656439
- [Background] Kimmig R, Aktas B, Buderath P, Wimberger P, Iannaccone A, Heubner M. Definition of compartment-based radical surgery in uterine cancer: modified radical hysterectomy in intermediate/high-risk endometrial cancer using peritoneal mesometrial resection (PMMR) by M Hockel translated to robotic surgery. World J Surg Oncol. 2013 Aug 16;11:198. doi: 10.1186/1477-7819-11-198. PMID 23947937
- [Background] Hockel M. Long-term experience with (laterally) extended endopelvic resection (LEER) in relapsed pelvic malignancies. Curr Oncol Rep. 2015 Mar;17(3):435. doi: 10.1007/s11912-014-0435-8. PMID 25687807
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Chi DS, Franklin CC, Levine DA, Akselrod F, Sabbatini P, Jarnagin WR, DeMatteo R, Poynor EA, Abu-Rustum NR, Barakat RR. Improved optimal cytoreduction rates for stages IIIC and IV epithelial ovarian, fallopian tube, and primary peritoneal cancer: a change in surgical approach. Gynecol Oncol. 2004 Sep;94(3):650-4. doi: 10.1016/j.ygyno.2004.01.029. PMID 15350354
- [Derived] Park SJ, Mun J, Lee S, Luo Y, Chung HH, Kim JW, Park NH, Song YS, Kim HS. Laterally Extended Endopelvic Resection Versus Chemo or Targeted Therapy Alone for Pelvic Sidewall Recurrence of Cervical Cancer. Front Oncol. 2021 May 25;11:683441. doi: 10.3389/fonc.2021.683441. eCollection 2021. PMID 34113571